CLINICAL TRIAL: NCT01309568
Title: "Quidel Reader Influenza A + B Test 510(k) and CLIA Waiver Field Study"
Status: Completed | Type: Observational
Sponsor: Quidel Corporation (Industry)
Responsible Party: John D. Tamerius, PhD, Sr. V.P. Clinical/Regulatory, Quidel Corporation
Other Study IDs: CS-0138-01-A
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Leftover nasal mucus placed in viral transport media will be retained after culture for possible RT-PCR.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Investigational testing: Pending the outcome of culture, the subject may be treated with an approved antiviral medication at the doctors discretion.

SUMMARY:
The objective of this study is to demonstrate the clinical performance of the Quidel Reader Influenza A+B test and Quidel Reader with the following sample types: nasal swab, nasopharyngeal swab, and nasopharyngeal aspirate/wash. Clinical performance will be based on comparison of Quidel Reader Influenza A+B results to cell culture at a Central Reference or Alternative Laboratory.

DETAILED DESCRIPTION:
A sufficient number of subjects will be enrolled to achieve a required minimum of cell culture-positive specimens for each sample type, nasal swab, nasopharyngeal swab, and nasopharyngeal aspirate/wash.

* The 510(k) study will include combined results from all sites and require the following for all three sample types: a minimum of 50 fresh positive results for influenza A, and 30 fresh positive results for influenza B.
* The CLIA Waiver submission will include combined results from all sites for a total of 120 positive specimens for both influenza A and influenza B. The nasal swab will be the primary sample type planned for the CLIA Waiver submission. However, depending upon the prevalence of influenza, nasopharyngeal swab and/or nasopharyngeal aspirate/wash may also be submitted for CLIA Waiver.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, of all ages (assuming appropriate consent is obtained).
2. Must currently be exhibiting symptoms characteristic of influenza-like-illness (ILI).

For example:

1. Fever, ≥ 38º C (100º F), either at the time of the visit or onset within the past two (2) days.
2. Nasal congestion
3. Rhinorrhea
4. Sore throat
5. Cough
6. Headache
7. Myalgia
8. Malaise

Exclusion Criteria:

1. Has undergone treatment with anti-influenza antivirals within the previous 7 days, including, for example, one or more of the following, but not be limited to Amantadine, Rimantadine, Ribavirin, Oseltamivir, Zanamivir or any other antiviral currently available in these classes.
2. Has been vaccinated by means of an influenza nasal spray/mist vaccine within the previous 7 days.
3. Unable to understand and consent to participation; for minors this includes parent or legal guardian.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects current exhibiting influenza like illness.
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Diagnosis of infection with influenza | 15 minutes
  Accurate diagnosis of infection with influenza A or influenza B confirmed by culture

CONTACTS AND LOCATIONS:
Overall Officials: John D Tamerius, PhD, Study Director — Quidel Corporation
Locations (16):
- United States (16):
  - La Costa Pediatrics, Carlsbad, California
  - Santo Nino Medical Clinic, Panorama City, California
  - La Jolla Pediatrics, San Diego, California
  - Complete Family Care, Northglenn, Colorado
  - Adriana Castro, MD, Miami, Florida
  - Teena Hughes, MD, Tampa, Florida
  - DuPage Family Medicine, Naperville, Illinois
  - Paul Janson, MD, Florence, Kentucky
  - Paul McLaughlin, MD, Mount Sterling, Kentucky
  - Kamakshi Neelkantan, MD, Edgewood, Maryland
  - Priority Care Pediatrics, Kansas City, Missouri
  - Robert Farron, DO, Far Rockaway, New York
  - Twelve Corners Pediatrics, Rochester, New York
  - Montrose Family Practice, Akron, Ohio
  - Norristown Family Physicians, Norristown, Pennsylvania
  - Dell's Children's Medical Center, Austin, Texas